CLINICAL TRIAL: NCT04348708
Title: An Open-Label, Long-Term Follow Up Study of Safety and Efficacy in PKU Subjects With PAH Deficiency Previously Administered HMI 102
Brief Title: Long-Term Follow Up Study of Subjects Previously Administered HMI 102
Status: Enrolling by invitation | Type: Observational
Sponsor: Homology Medicines, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: HMI-102-102
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Phenylketonuria; PAH Deficiency
Keywords: PKU; Phenylketonuria; PAH Deficiency; Phenylalanine; Adeno Associated Virus; AAVHSC15
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Neutralizing AAV antibody, AAV antibody (IgG), Anti-PAH antibody, Vector DNA in blood, Vector DNA in body fluids, Serum Chemistry, Hematology
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Dose Level Cohort 1: Dose Level 1 of HMI-102 delivered intravenously one time
  Interventions: Genetic: HMI-102
- Dose Level Cohort 2: Dose Level 2 of HMI-102 delivered intravenously one time
  Interventions: Genetic: HMI-102
- Dose Level Cohort 3: Dose Level 3 of HMI-102 delivered intravenously one time
  Interventions: Genetic: HMI-102

INTERVENTIONS:
Genetic: HMI-102 — HMI-102 is an AAVHSC15 vector containing a functional copy of the human PAH gene

SUMMARY:
An Open-Label, Long-Term Follow Up Study of Safety and Efficacy in PKU Subjects with PAH Deficiency Previously Administered HMI 102

DETAILED DESCRIPTION:
This Long-Term Follow Up Study will evaluate the safety and efficacy of PKU Subjects with PAH Deficiency Previously Administered HMI 102. Subjects will have already received a single dose of HMI-102 administered intravenously

ELIGIBILITY:
Inclusion Criteria:

* Subject was previously administered HMI 102.
* Subject is able to understand the purpose and risks of the study and is willing to provide informed consent.
* Subject is able to comply with all study procedures and long-term follow-up.

Exclusion Criteria:

* Participation in the study is not in the subject's best interest, in the opinion of the Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects with PAH Deficiency who were previously administered HMI-102
Sampling Method: Non-Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2020-08-19 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events of special interest (AESIs) and serious adverse events (SAEs) related to HMI 102 | Baseline to year 5
  Subjects with at least one AESI or SAE

SECONDARY OUTCOMES:
Plasma Phe Concentration | Baseline to year 5
  Plasma phenylalanine (Phe) concentration at each time point during the study
Phe-restricted diet | Baseline to year 5
  Incidence of subjects with a Phe-restricted diet
Phenylketonuria Quality of Life Questionnaire (PKU-QOL | Baseline to year 5
  Quality of life (QOL), as assessed using the Phenylketonuria-QOL (PKU-QOL) questionnaire
Protein intake | Baseline to year 5
  Protein intake relative to Phe concentration at each time point during the study

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York